CLINICAL TRIAL: NCT00797030
Title: Topical Cyclosporine for the Treatment of Dry Eye in Patients Infected With the Human Immunodeficiency Virus
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Rodrigo de Pinho Paes Barreto, MD, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: dry eye
Record Dates: First submitted 2008-11-21; First posted 2008-11-24 (Estimated); Last update posted 2008-11-24 (Estimated); Status verified 2008-11

CONDITIONS: Dry Eye Syndromes; HIV Seropositivity
Keywords: dry eye syndromes; keratoconjuntivitis sicca / drug therapy; cyclosporine; ophthalmic solutions; HIV seropositivity
MeSH Terms: conditions — Dry Eye Syndromes; HIV Seropositivity | interventions — Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Ten HIV-positive-patients with dry eye diagnosis received sodium carboxymethylcellulose 0.5% drops (one drop 4 times per day) and topical cyclosporine 0.05% (one drop twice a day) for six months.
  Interventions: Drug: cyclosporine and sodium carboximethycellulose
- 2 (Other): Ten HIV-positive-patients with dry eye received sodium carboximethylcelullose 0.5% (1 drop 4 times per day) during six months
  Interventions: Drug: sodium carboximethycellulose

INTERVENTIONS:
Drug: cyclosporine and sodium carboximethycellulose — Ten HIV-positive patients with dry eye received sodium carboximethylcellulose 0.5% (one drop 4 times per day) and topical cyclosporine 0.05% (one drop twice a day) during six months
  Arms: 1
Drug: sodium carboximethycellulose — Ten HIV-positive patients with dry eye received sodium carboximethycellulose (1 drop 4 times per day) during six months
  Arms: 2

SUMMARY:
This study evaluates the use of topical cyclosporine 0.05% and sodium carboxymethylcellulose 0.5% for the treatment of dry eye disease in patients infected with the human immunodeficiency virus.

Twenty HIV-positive-patients were selected from the Department of Infectious Diseases of the Federal University of Rio de Janeiro Hospital. Dry eye diagnosis was based on a dry eye questionnaire (Ocular Surface Disease Index - OSDI®), Schirmer I Test, break up time and 1% rose bengal staining of the ocular surface. The patients were divided into two groups with ten patients. Group I received sodium carboxymethylcellulose 0.5% drops and group II received sodium carboxymethylcellulose 0,5% drops and topical cyclosporine 0.05% for six months.

ELIGIBILITY:
Inclusion Criteria:

* HIV seropositivity
* Dry eye diagnosis

Exclusion Criteria:

* Hepatitis B infection
* Hepatitis C infection
* Menopause
* Rheumatic diseases
* Contact lens wear
* Beta-blocker eye drops
* Blepharitis
* Use of medications associated with dry eye (diuretics, antidepressive agents, beta-blockers)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2006-10; Primary Completion 2008-07 (Estimated); Study Completion 2008-11 (Estimated)

PRIMARY OUTCOMES:
Dry eye diagnosis was based on a dry eye questionnaire (OSDI), Shirmer I Test, BUT and 1% rose bengal staining of the ocular surface. The same tests were performed at the end of the treatment to verify the improvement of the subjects. | six months

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo P Barreto, Masters, Principal Investigator — Universidade Federal do Rio de Janeiro
Locations (1):
- Universidade Federal do Rio de Janeiro, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Background] Cunningham ET Jr, Margolis TP. Ocular manifestations of HIV infection. N Engl J Med. 1998 Jul 23;339(4):236-44. doi: 10.1056/NEJM199807233390406. No abstract available. PMID 9673303
- [Background] Kordossis T, Paikos S, Aroni K, Kitsanta P, Dimitrakopoulos A, Kavouklis E, Alevizou V, Kyriaki P, Skopouli FN, Moutsopoulos HM. Prevalence of Sjogren's-like syndrome in a cohort of HIV-1-positive patients: descriptive pathology and immunopathology. Br J Rheumatol. 1998 Jun;37(6):691-5. doi: 10.1093/rheumatology/37.6.691. PMID 9667626
- [Background] DeCarlo DK, Penner SL, Schamerloh RJ, Fullard RJ. Dry eye among males infected with the human immunodeficiency virus. J Am Optom Assoc. 1995 Sep;66(9):533-8. PMID 7490413
- [Background] Geier SA, Libera S, Klauss V, Goebel FD. Sicca syndrome in patients infected with the human immunodeficiency virus. Ophthalmology. 1995 Sep;102(9):1319-24. doi: 10.1016/s0161-6420(95)30868-8. PMID 9097769
- [Background] Lucca JA, Kung JS, Farris RL. Keratoconjunctivitis sicca in female patients infected with human immunodeficiency virus. CLAO J. 1994 Jan;20(1):49-51. PMID 8149575
- [Background] Lucca JA, Kung JS, Farris RL. Keratoconjunctivitis sicca in HIV-1 infected female patients. Adv Exp Med Biol. 1994;350:521-3. doi: 10.1007/978-1-4615-2417-5_87. No abstract available. PMID 8030528
- [Background] Lucca JA, Farris RL, Bielory L, Caputo AR. Keratoconjunctivitis sicca in male patients infected with human immunodeficiency virus type 1. Ophthalmology. 1990 Aug;97(8):1008-10. doi: 10.1016/s0161-6420(90)32472-7. PMID 2402409
- [Background] Lemp MA. Report of the National Eye Institute/Industry workshop on Clinical Trials in Dry Eyes. CLAO J. 1995 Oct;21(4):221-32. No abstract available. PMID 8565190